CLINICAL TRIAL: NCT04117659
Title: Right Ventricular Function After Withdrawal of Phosphodiesterase-5 Inhibitors in Left Ventricular Assist Device Recipients
Brief Title: Phosphodiesterase-5-inhibitors for Right Heart Failure After Left Ventricular Assist Device Implantation
Acronym: PIVAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maria Papathanasiou, Principal Investigator, Cardiologist, University Hospital, Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 177923
Record Dates: First submitted 2019-08-22; First posted 2019-10-07 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Phosphodiesterase Inhibitor Adverse Reaction; Right-Sided Heart Failure
Keywords: Left ventricular assist device; postoperative right heart failure
MeSH Terms: conditions — Heart Failure | interventions — Phosphodiesterase 5 Inhibitors

STUDY DESIGN:
Intervention Model Description: withdrawal of a pharmacologic therapy in pre-treated patients without control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phosphodiesterase-5 inhibitor withdrawal (Experimental): In this single arm pretreatment with an oral phosphodiesterase-5 inhibitor will be discontinued
  Interventions: Other: withdrawal of oral medication (phosphodiesterase-5 inhibitor) in pretreated patients

INTERVENTIONS:
Other: withdrawal of oral medication (phosphodiesterase-5 inhibitor) in pretreated patients — discontinuation of the oral medication with a phosphodiesterase-5 inhibitor

SUMMARY:
Refractory right heart failure is common during the postoperative period after left ventricular assist device implantation. Oral phosphodiesterase-5 inhibitors are oft initiated in order to facilitate weaning from the intravenous inotropic substances. following this period many patients continue to receive the same medication in the long term, despite missing data on its therapeutic effect on right ventricular function.We hypothesise that beyond the acute postoperative period no additional benefit from the phosphodiesterase-5 inhibitors exists. The aim of the study is a detailed clinical and echocardiographic assessment of the right ventricular function after discontinuation of the medication in patients pretreated for at least one month after receiving left ventricular assist device.

DETAILED DESCRIPTION:
The study aims to assess clinical and echocardiographic measures of right ventricular function before and after discontinuation of the oral phosphodiesterase-5 inhibitor in patients on left ventricular device support. At baseline and after discontinuation of the medication patients will receive a clinical examination and New York Heart Association Classification, echocardiographic assessment of right ventricular function, cardiopulmonary exercise testing, 6 minute walking test and assessment of quality of life. The primary outcome is the change of the quantitative echocardiographic parameters of right ventricular function at follow-up. Secondarily, we aim to assess the change in cardiopulmonary exercise capacity, the 6-minute walking distance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 y.o.
* clinically stable, ambulatory heart failure patients on left ventricular assist device support
* implantation > 1 month before inclusion in the study
* uninterrupted therapy with an oral phosphodiesterase-5 inhibitor initiated during the early postoperativ period due to right heart failure

Exclusion Criteria:

* unable to provide written informed consent
* refusal to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in right ventricular global longitudinal strain | 4 weeks after discontinuation of phosphodiesterase-5 inhibitors
  Change in right ventricular function from baseline as assessed by global longitudinal strain of the right ventricle on transthoracic echocardiography

SECONDARY OUTCOMES:
Change from baseline in peak oxygen uptake rate | 4 weeks after discontinuation of phosphodiesterase-5 inhibitors
  Change from baseline in functional status as estimated by peak oxygen uptake rate in cardiopulmonary exercise testing
Change from baseline in 6-minute walking distance | 4 weeks after discontinuation of phosphodiesterase-5 inhibitors
  Change from baseline in walking distance assessed by 6-minute walking test
Change from baseline in the total score of quality of life calculated with the Kansas City Cardiomyopathy Questionnaire | 4 weeks after discontinuation of phosphodiesterase-5 inhibitors
  Change from baseline in the total score calculated with the Kansas City Cardiomyopathy Questionnaire (range between 0 and 100, higher value indicates worse status of quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Papathanasiou, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trachte AL, Lobato EB, Urdaneta F, Hess PJ, Klodell CT, Martin TD, Staples ED, Beaver TM. Oral sildenafil reduces pulmonary hypertension after cardiac surgery. Ann Thorac Surg. 2005 Jan;79(1):194-7; discussion 194-7. doi: 10.1016/j.athoracsur.2004.06.086. PMID 15620942
- [Background] Kormos RL, Teuteberg JJ, Pagani FD, Russell SD, John R, Miller LW, Massey T, Milano CA, Moazami N, Sundareswaran KS, Farrar DJ; HeartMate II Clinical Investigators. Right ventricular failure in patients with the HeartMate II continuous-flow left ventricular assist device: incidence, risk factors, and effect on outcomes. J Thorac Cardiovasc Surg. 2010 May;139(5):1316-24. doi: 10.1016/j.jtcvs.2009.11.020. Epub 2010 Feb 4. PMID 20132950
- [Background] Hamdan R, Mansour H, Nassar P, Saab M. Prevention of right heart failure after left ventricular assist device implantation by phosphodiesterase 5 inhibitor. Artif Organs. 2014 Nov;38(11):963-7. doi: 10.1111/aor.12277. Epub 2014 Apr 2. PMID 24689700
- [Background] Baker WL, Radojevic J, Gluck JA. Systematic Review of Phosphodiesterase-5 Inhibitor Use in Right Ventricular Failure Following Left Ventricular Assist Device Implantation. Artif Organs. 2016 Feb;40(2):123-8. doi: 10.1111/aor.12518. Epub 2015 Jun 4. PMID 26043796
- [Background] Klodell CT Jr, Morey TE, Lobato EB, Aranda JM Jr, Staples ED, Schofield RS, Hess PJ, Martin TD, Beaver TM. Effect of sildenafil on pulmonary artery pressure, systemic pressure, and nitric oxide utilization in patients with left ventricular assist devices. Ann Thorac Surg. 2007 Jan;83(1):68-71; discussion 71. doi: 10.1016/j.athoracsur.2006.08.051. PMID 17184632
- [Background] Tedford RJ, Hemnes AR, Russell SD, Wittstein IS, Mahmud M, Zaiman AL, Mathai SC, Thiemann DR, Hassoun PM, Girgis RE, Orens JB, Shah AS, Yuh D, Conte JV, Champion HC. PDE5A inhibitor treatment of persistent pulmonary hypertension after mechanical circulatory support. Circ Heart Fail. 2008 Nov;1(4):213-9. doi: 10.1161/CIRCHEARTFAILURE.108.796789. PMID 19808294
- [Background] Feldman D, Pamboukian SV, Teuteberg JJ, Birks E, Lietz K, Moore SA, Morgan JA, Arabia F, Bauman ME, Buchholz HW, Deng M, Dickstein ML, El-Banayosy A, Elliot T, Goldstein DJ, Grady KL, Jones K, Hryniewicz K, John R, Kaan A, Kusne S, Loebe M, Massicotte MP, Moazami N, Mohacsi P, Mooney M, Nelson T, Pagani F, Perry W, Potapov EV, Eduardo Rame J, Russell SD, Sorensen EN, Sun B, Strueber M, Mangi AA, Petty MG, Rogers J; International Society for Heart and Lung Transplantation. The 2013 International Society for Heart and Lung Transplantation Guidelines for mechanical circulatory support: executive summary. J Heart Lung Transplant. 2013 Feb;32(2):157-87. doi: 10.1016/j.healun.2012.09.013. No abstract available. PMID 23352391